CLINICAL TRIAL: NCT04021693
Title: Does Improved Access to a Portable Ultrasound Device Improve Trainee Learning With Point-of-care Ultrasonography: A Randomized Trial
Brief Title: Learning Outcomes With Point-of-Care Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andre Kumar, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 42094
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Ultrasound
Keywords: Medical Education

STUDY DESIGN:
Intervention Model Description: Intern physicians were randomized 1:1 to receive personal access to a handheld ultrasound device vs. no device. The groups did not cross over in which intervention they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handheld Ultrasound Devices (Experimental)
  Interventions: Other: Handheld Ultrasound Devices
- No Handheld Ultrasound Devices (No Intervention)

INTERVENTIONS:
Other: Handheld Ultrasound Devices — Interns in the handheld ultrasound device arm shall carry a personal handheld ultrasound device to be used for self-directed learning
  Arms: Handheld Ultrasound Devices

SUMMARY:
Point-of care-ultrasonography has the potential to transform healthcare delivery through its diagnostic and therapeutic utility. Its use has become more widespread across a variety of clinical settings as more investigations have demonstrated its impact on patient care. This includes the use of point-of-care ultrasound by trainees, who are now utilizing this technology as part of their diagnostic assessments of patients. However, there are few studies that examine how efficiently trainees can learn point-of-care ultrasound and which training methods are more effective. The primary objective of this study is to assess whether handheld ultrasound devices, along with a year-long lecture series, improve internal medicine interns' knowledge and image interpretation skills with point-of-care ultrasound. Participants shall be randomized to receive personal access to handheld ultrasound devices to be used for learning vs. no personal access. The primary outcome will assess their interpretive ability with ultrasound images/videos. Secondary outcomes will include rates of device usage and lecture attendance.

ELIGIBILITY:
Inclusion Criteria:

* Internal Medicine Intern Physicians at Stanford University

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Mean Percent Correct On Image Assessments at 1 year | 1 year
  Image assessments will include videos and photographs of ultrasound images that will require the intern to interpret the image.

SECONDARY OUTCOMES:
Mean Reported Device Usage Rates at 1 year | 1 year
  Self-reported usage rates of the ultrasound devices per week by the interns
Mean Lecture Attendance at 1 year | 1 year
  Mean Lecture Attendance per Study Arm

CONTACTS AND LOCATIONS:
Overall Officials: Andre D Kumar, MD, MEd, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Kugler J, Jensen T. Evaluation of Trainee Competency with Point-of-Care Ultrasonography (POCUS): a Conceptual Framework and Review of Existing Assessments. J Gen Intern Med. 2019 Jun;34(6):1025-1031. doi: 10.1007/s11606-019-04945-4. PMID 30924088
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104